CLINICAL TRIAL: NCT06529783
Title: Effectiveness of Ultrasound-Guided Percutaneous Neuromodulation (UG-PNM) on the Superior Gluteal Nerve in Patients With Greater Trochanteric Pain Syndrome (GTPS): A Pilot Study
Brief Title: Ultrasound-Guided Percutaneous Neuromodulation on the Superior Gluteal Nerve in Patients With Greater Trochanteric Pain Syndrome: A Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Dr. Pablo Herrero Gallego, Principal Investigator, Universidad de Zaragoza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NMP-e.STM
Record Dates: First submitted 2024-07-26; First posted 2024-07-31 (Actual); Last update posted 2025-06-02 (Actual); Status verified 2025-05

CONDITIONS: Greater Trochanteric Pain Syndrome
Keywords: Neromodulation; Percutaneous; ultrasound; superior gluteal nerve
MeSH Terms: interventions — Extracorporeal Shockwave Therapy; Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shockwave Therapy + Therapeutic Exercises (Active Comparator): Patients on this group receive two interventions based on Shockwave Therapy and Therapeutic Exercises
  Interventions: Other: Shockwave Therapy; Other: Therapeutic Exercises
- Shockwave Therapy + Therapeutic Exercises + US-Guided percutaneous neuromodulation (Experimental): Patients on this group receive both interventions previously described and ultrasound-guided percuteneous neuromodulation is added.
  Interventions: Other: Shockwave Therapy; Other: Therapeutic Exercises; Other: Ultrasound-Guided Percutaneous Neuromodulation:

INTERVENTIONS:
Other: Shockwave Therapy — The proposed model for radial shockwave therapy at Clínica Osteopática Dr. David Ponce is the DolorClast® by EMS, made in Nyon, Switzerland. Treatment parameters include 2500 impulses, 0.2 mJ/mm² energy density, and 15 pulses per second, using a 15 mm diameter applicator with ultrasound gel applied to the treatment area. The patient will be positioned laterally on the table with specific leg positions to ensure comfort and effectiveness.
Other: Therapeutic Exercises — The exercise protocol was followed daily, with continuous physiotherapist supervision to ensure correct execution and avoid improper postures. The protocol includes four exercises: bilateral low-load supine abduction, unilateral isometric hip abduction in medial rotation, hip abduction with sliding, and bilateral supported glute bridge. A maximum of 4/10 on the VAS pain scale is allowed during exercise; exceeding this threshold means skipping exercises for that day.
Other: Ultrasound-Guided Percutaneous Neuromodulation: — This technique was applied only to the experimental group before shockwave therapy. An ultrasound-guided approach to the superior gluteal nerve used a 7-12 MHz linear probe from Esaote MyLab™Alpha and Physio Invasiva® equipment. The needle length varied with patient anatomy, with a typical safety reference from 0.30 x 60 to 0.35 x 70 mm. A biphasic current with 10 Hz frequency and 240 μs pulse width was used, with intensity adjusted for a visible but non-painful motor response, following the 10-10-10 protocol.
  To locate the superior gluteal nerve, a longitudinal scan of the lateral iliac crest identified the nerve between the gluteus minimus and medius. The procedure used a short-axis approach at 80º to target the nerve's perineurium, with the area disinfected with chlorhexidine before needle insertion.
  Arms: Shockwave Therapy + Therapeutic Exercises + US-Guided percutaneous neuromodulation

SUMMARY:
Greater Trochanteric Pain Syndrome (GTPS) predominantly affects women, with an annual incidence of 1.8 to 5.6 per 1000 individuals and a prevalence ratio of 4:1 compared to men. It is characterized by lateral pain in the greater trochanter region, particularly during palpation, prolonged sitting, and physical activity. Conservative treatments, such as radial shockwave therapy and therapeutic exercises, are effective but slow, and some patients eventually require surgery.

Ultrasound-guided percutaneous neuromodulation, targeting the superior gluteal nerve, has emerged as a promising alternative to improve GTPS outcomes. This technique aims to normalize motor response and reduce pain more rapidly than conventional therapies. Integrating neuromodulation could accelerate recovery, enhancing both pain relief and tendon functionality. This study aims to explore the effectiveness of this technique as an adjunct to conventional treatments, aiming for faster symptom improvement and better long-term adherence.

DETAILED DESCRIPTION:
Greater Trochanteric Pain Syndrome (GTPS) is a condition primarily affecting women, with an annual incidence ranging from 1.8 to 5.6 per 1000 individuals and a prevalence ratio of 4:1 compared to men. Formerly known as trochanteric bursitis, this syndrome is characterized by lateral pain in the region of the greater trochanter, particularly manifesting during palpation, prolonged sitting, and physical activity. The primary cause of GTPS is attributed to repetitive friction between the greater trochanter and the iliotibial band, resulting in gluteus medius or minimus tendinopathy, as well as other associated conditions such as trochanteric bursitis and iliotibial band syndrome.

Conservative treatment is the first-line approach for GTPS, with radial shockwave therapy and therapeutic exercises demonstrating long-term efficacy. However, a percentage of patients require surgical intervention due to a lack of response to conservative treatments.

Ultrasound-guided percutaneous neuromodulation, a technique utilizing electrical stimulation via a needle guided by ultrasound, has emerged as a potential alternative to improve therapeutic outcomes for GTPS. In this study, this technique targets the superior gluteal nerve, which innervates the gluteus medius, minimus, and tensor fasciae latae, with the aim of normalizing motor response and reducing pain. Neuromodulation could provide a faster improvement in symptoms and motor patterns compared to conventional therapies, which require prolonged periods to be effective.

Given that current treatments for GTPS, such as shockwave therapy and therapeutic exercises, are effective but slow in progress, the integration of percutaneous neuromodulation could accelerate patient recovery, improving both pain relief and mechanical functionality of the tendon. This combined approach has the potential not only to optimize clinical outcomes but also to reduce the need for surgical interventions in GTPS patients.

In summary, this study proposes to explore the effectiveness of superior gluteal nerve neuromodulation as an adjunct to conventional treatments for GTPS. The research aims to demonstrate whether this technique can significantly expedite pain reduction and motor pattern improvement, thereby enhancing long-term treatment adherence and tolerance.

ELIGIBILITY:
Inclusion Criteria:

* Suffering from Greater Trochanteric Pain Syndrome (GTPS).
* Experiencing local pain upon palpation of the greater trochanter area.
* Having pain in the greater trochanter region lasting more than three months, indicating chronicity.
* Being over 18 years of age.
* Experiencing pain when bearing weight on the affected trochanter.
* Having pain that impairs the functionality of resisted hip abduction.

Exclusion Criteria:

* Radiological evidence of pathology in the hip or knee joints.
* Blood coagulation disorders.
* Use of oral anticoagulants.
* Presence of infections.
* History of disc or hip surgery.
* Presence of dysplasia, deformities, or sciatica.
* History of vascular, neurological, or neoplastic diseases.
* Specific contraindications for ultrasound-guided percutaneous neuromodulation (UG-PNM): belenophobia, pregnancy, pacemakers, epilepsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-26 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Functional capacity | This variable is measured five times, corresponding with the five participant visits (day 1, week 4, week 8, week 16, and year 1).
  Functionality will be assessed using the Visa-G questionnaire, which consists of 8 questions divided into three main aspects: pain, function, and activity. The first 7 questions score up to 10 points each, while question 8 has a maximum score of 30. An asymptomatic person would score a total of 100 points; thus, a lower score indicates greater disability severity.

SECONDARY OUTCOMES:
Pain on the Day Prior to the Visit | This variable is collected on five occasions, coinciding with the five participant visits (day 1, week 4, week 8, week 16, and year 1)
  Pain is measured using the Visual Analog Scale (VAS).
Pain on Palpation of the Greater Trochanter | day 1, week 4, week 8, week 16, and year 1
  Pain on palpation, performed by the physiotherapist, is also measured using the VAS
Hip Abductor Muscle Strength | day 1, week 4, week 8, week 16, and year 1
  Strength is measured using an Active Force 2 dynamometer
Adverse Effects | day 1, week 4, week 8, week 16, and year 1
  Adverse effects for this study include pain during the treatment session, pain after the session, inflammation and/or redness in the treated area, bruising in the treated region, dizziness, muscle fatigue, numbness, and drowsiness. These are assessed through the participant's oral reports.
Adherence to the Therapeutic Exercise Protocol | day 1, week 4, week 8, week 16, and year 1
  Adherence is assessed by asking the patient in each session if they are following the protocol correctly, with an emphasis on honesty to ensure accurate recording of adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Herrero, Physiotherapist, Study Director — Universidad de Zaragoza
Locations (1):
- University of Zaragoza, Zaragoza, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared on a reasonable request contacting with the main author once data has been published.
  Anyway, Individual participant data (IPD) will be shared with other researchers in accordance with data sharing protocols and participant consent, ensuring confidentiality and ethical considerations are maintained.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Once research has been published
Access Criteria: Study protocol will be publish in a scientific journal